CLINICAL TRIAL: NCT03101371
Title: Reducing Urinary Tract Infection Rates Using a Controlled Aseptic Protocol for Catheter Insertion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-1096
Record Dates: First submitted 2017-03-30; First posted 2017-04-05 (Actual); Results first posted 2020-02-18 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Urinary Tract Infections; Catheter Infection; Catheter-Related Infections
MeSH Terms: conditions — Urinary Tract Infections; Catheter-Related Infections | interventions — Catheterization; Povidone-Iodine

STUDY DESIGN:
Intervention Model Description: Patients with normal urinary analysis (UA) pre-surgery will be randomized 1:1 to one of two arms prior to surgery:
  1. Aseptic protocol for catheter insertion using Povidone Iodine treated catheter and maintaining plastic sleeve on catheter or
  2. Standard of care (SOC) catheter insertion in which catheter is inserted right out of package/non-treated catheter.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care catheter insertion (Active Comparator): Standard of care catheter insertion in which catheter is inserted right out of package/non-treated catheter.
  Interventions: Procedure: Standard of care catheter insertion
- Aseptic protocol for catheter insertion (Experimental): Aseptic protocol for catheter insertion using Povidone Iodine treated catheter and maintaining plastic sleeve on catheter
  Interventions: Drug: Catheter insertion with Povidone Iodine

INTERVENTIONS:
Drug: Catheter insertion with Povidone Iodine — The catheter will be treated with Povidone Iodine prior to insertion.
  Other Names: Aseptic protocol for catheter insertion using Povidone Iodine treated catheter
  Arms: Aseptic protocol for catheter insertion
Procedure: Standard of care catheter insertion — Catheter inserted right out of package.
  Arms: Standard of care catheter insertion

SUMMARY:
Urinary Tract Infection (UTI) complications following catheter use in surgical patients remains high. Using an aseptic protocol has been shown to drastically reduce UTI incidence by 50%. Reducing UTIs will prevent extended hospital stays, readmission, and antibiotic use associated with this complication and improve cost-effectiveness of care. The investigators hypothesize that they can reduce the incidence of UTIs after catheter placement with the implementation of a Quality Improvement (QI) protocol to prevent excess exposure to the environment exposure of the catheter before, during and after insertion.

ELIGIBILITY:
Inclusion Criteria:

1. women 18-89 years of age
2. admitted for surgery lasting >1 hour and requiring urinary catheter,
3. have normal urine analysis within 24 hours pre-surgery, and
4. able to provide informed consent.

Exclusion Criteria:

1. currently on dialysis,
2. chronic urinary infection,
3. hyperthyroidism,
4. current infection,
5. a history of allergy or sensitivity to iodine.
6. women who are pregnant or breast feeding
7. men due to their lower incidence of UTIs compared to the female population.

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 99 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saketh Guntupalli, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A single-site randomized controlled trial, conducted at the University of Colorado Hospital, enrolled women beginning October 2017 and ended February 2019.
Groups:
- Standard of Care Protocol Catheter Insertion: Standard of care catheter insertion in which catheter is inserted right out of package/non-treated catheter.
  Standard of care catheter insertion: Catheter inserted right out of package.
Period: Overall Study
Arm/Group | Standard of Care Protocol Catheter Insertion | Aseptic Protocol for Catheter Insertion
Started | 48 | 51
Completed | 45 | 45
Not Completed | 3 | 6
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 1 | 4
Not completed — Did not meet eligibility criteria | 2 | 1

BASELINE CHARACTERISTICS:
Population: 99 participants were randomized, however, 9 participants were excluded from analsysis due to early discontinuation for not meeting eligibility criteria (n=3), provider discretion (n=1), and lost to follow-up (n=5).
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Protocol Catheter Insertion | Aseptic Protocol for Catheter Insertion | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (13.37) | 56.5 (14.27) | 56.2 (13.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 45 | 90
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnic group: White Non-Hispanic | 40 | 36 | 76
  Race/ethnic group: Hispanic | 2 | 6 | 8
  Race/ethnic group: American Indian or Alaskan Native | 1 | 0 | 1
  Race/ethnic group: African American | 1 | 1 | 2
  Race/ethnic group: Asian | 1 | 2 | 3
Menopause status [Count of Participants; unit: Participants]
  Pre-menopausal | 15 | 15 | 30
  Post-menopausal | 30 | 30 | 60
Smoking status [Count of Participants; unit: Participants]
  Current | 5 | 6 | 11
  Former | 12 | 17 | 29
  Never | 28 | 22 | 50
Diabetes [Count of Participants; unit: Participants] | 4 | 6 | 10
Hypertension [Count of Participants; unit: Participants] | 16 | 18 | 34
Cancer Diagnosis [Count of Participants; unit: Participants]
  Uterine Cancer | 10 | 10 | 20
  Ovarian Cancer | 26 | 24 | 50
  Cervical | 2 | 2 | 4
  Benign | 5 | 8 | 13
  Other | 2 | 1 | 3
Primary Surgery [Count of Participants; unit: Participants]
  Total Abdominal Hysterectomy +/- BSO/USO | 23 | 28 | 51
  Radical Hysterectomy | 2 | 0 | 2
  Bowel resection | 4 | 2 | 6
  Omentectomy | 6 | 4 | 10
  Bilateral/unilateral salpingo-oophorectomy | 3 | 5 | 8
  Lymph Node Dissection | 1 | 0 | 1
  Other | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Catheter Associated Urinary Tract Infection (CAUTI)
Description: Participants were monitored for up to 14 days. This was assessed with a rapid urine analysis (UA) test. A urinary tract infection was defined as >10^5 bacterial colony forming units per ML on urine culture regardless of symptoms. This is the number of participants who had at least one CAUTI during the time of observation.
Time Frame: Within 14 +/- 2 days post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Protocol Catheter Insertion | Aseptic Protocol for Catheter Insertion
Number analyzed (Participants) | 45 | 45
Participants | 7 | 6

2. Secondary Outcome: Number of Participants Who Received the "Fill and Pull" Versus the "Pull and Void" Method of Catheter Discontinuation
Description: Participants were monitored for up to 2 weeks. This is the number of participants who received one method versus the other for catheter discontinuation.
Time Frame: Day 14 (+/- 2 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Protocol Catheter Insertion | Aseptic Protocol for Catheter Insertion
Number analyzed (Participants) | 45 | 45
Participants
  Fill and pull | 38 | 40
  Pull and void | 7 | 5

3. Secondary Outcome: Average Patient Satisfaction
Description: Participants were monitored at 2 weeks. This was assessed using a Likert scale questionnaire (1 = not at all satisfied, 10 = extremely satisfied). Average patient satisfaction with the catheter was assessed.
Time Frame: Day14 (+/- 2 days)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care Protocol Catheter Insertion | Aseptic Protocol for Catheter Insertion
Number analyzed (Participants) | 45 | 45
score on a scale | 8.17 (2.39) | 8.6 (2.04)

4. Secondary Outcome: Number of Participants With Extended Hospital Stay Due to a Urinary Tract Infection (UTI)
Description: Participants were monitored for up to 14 days. This is the number of participants who had a UTI in the hospital, extending their stay for more than seven days.
Time Frame: 14 days (+/- 2 days) from surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Protocol Catheter Insertion | Aseptic Protocol for Catheter Insertion
Number analyzed (Participants) | 45 | 45
Participants | 0 | 1

5. Secondary Outcome: Number of Participants With Closed Drainage System Disrupted During Placement of Catheter
Description: Participants were monitored post surgery until time of discharge. This is the number of participants who had the closed drainage system disrupted during placement of catheter for back fill of the bladder during surgery.
Time Frame: Day 1 post op
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Protocol Catheter Insertion | Aseptic Protocol for Catheter Insertion
Number analyzed (Participants) | 45 | 45
Participants | 42 | 42

6. Secondary Outcome: Number of Participants That Were Readmitted, Had Additional Clinic Visits or Went to the Emergency Department (ED) for Any Reason
Description: Participants were monitored up to two weeks. This is the number of participants who had at least one readmission or emergency room visit during the time of observation.
Time Frame: Day 14 (+/- 2 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Protocol Catheter Insertion | Aseptic Protocol for Catheter Insertion
Number analyzed (Participants) | 45 | 45
Participants | 0 | 1

7. Secondary Outcome: Number of Patients That Used Antibiotics at the Time of Surgery and Post-surgery
Description: Participants were monitored for up to 2 weeks. This is the number of participants that used any antibiotic during surgery and post-surgery.
Time Frame: Day 14 (+/- 2 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Protocol Catheter Insertion | Aseptic Protocol for Catheter Insertion
Number analyzed (Participants) | 45 | 45
Participants
  Cefazolin (1st gen cephalosporin)) | 36 | 39
  Cefoxitin Cefuroxime / Cefotetan (2nd gen cephalo | 5 | 0
  Metronidazole | 12 | 11
  Clindamycin | 5 | 6
  Doxycycline | 0 | 0
  Gentamicin | 3 | 6

ADVERSE EVENTS:
Time Frame: 14 days +/- 2 days post-surgery
Arm/Group | Standard of Care Protocol Catheter Insertion | Aseptic Protocol for Catheter Insertion
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 2/45 | 3/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care Protocol Catheter Insertion (N=45) | Aseptic Protocol for Catheter Insertion (N=45)
Catheter discomfort (Surgical and medical procedures) | 1 (1) | 1 (1)
Neutropenic fever (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/71/NCT03101371/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT03101371/ICF_001.pdf